CLINICAL TRIAL: NCT06617520
Title: Attitudes and Smoking Perceptions in the Real Environment
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Presbyterian Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ASPIRE; ST116745 (Other Grant/Funding Number: Presbyterian Health Foundation)
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tobacco flavor cigarillo (Experimental): A participant will use a tobacco flavored cigarillo at home for 7-days, as they wish, and then smoke it once in the laboratory
  Interventions: Other: Cigarillo flavor type
- Concept flavor cigarillo (Experimental): A participant will use a concept flavored cigarillo at home for 7-days, as they wish, and then smoke it once in the laboratory
  Interventions: Other: Cigarillo flavor type
- Characterizing flavor (Experimental): A participant will use a characterizing flavored cigarillo at home for 7-days, as they wish, and then smoke it once in the laboratory
  Interventions: Other: Cigarillo flavor type

INTERVENTIONS:
Other: Cigarillo flavor type — Participants will complete a within-subjects design that varies by cigarillo smoked: tobacco flavor, concept flavor, and characterizing flavor

SUMMARY:
This study will measure appeal and reinforcement for different flavored little cigars/cigarillos (LCCs) in young adults in the laboratory and at-home, via ecological momentary assessment (daily smart-phone surveys)

DETAILED DESCRIPTION:
Participants will attend 4 laboratory sessions that differ by cigarillo smoked: own brand and a then commercially available study cigarillo (Garcia y Vega game cigarillo) in tobacco flavor, concept flavor, and characterizing flavor. Consistent with our work and other's published work8-10, a baseline (BL) period will measure appeal to smoking one's usual brand cigarillo in their home environment for 7 days and then once in the laboratory (>12-hour abstinence), at the end of the 7 days. Participants will then undergo 3 experimental conditions (counterbalanced, within-subjects): (1) 7 days smoking a concept flavored study cigarillo; (2) 7 days smoking a characterizing flavored study cigarillo; and (3) 7 days smoking a tobacco flavored study cigarillo. Participants will be instructed to switch their usual brand cigarillo for the assigned study cigarillo for each 7-day period. Other tobacco use will be allowed during that time without specific instruction to model real-world behavior. On the last day of each 7-day period of "take home" use, abstinent participants (>12 hours) will smoke the assigned study cigarillo in the lab ad libitum, where subjective effects (e.g., satisfaction, craving reduction, psychological reward, throat hit), smoke exposure (CO boost), and behavior (e.g., number of puffs) will be assessed During each 7-day period of exposure, participants will complete assessments of cigarillo and other tobacco use and subjective effects to cigarillo use via once daily EMA.

ELIGIBILITY:
Inclusion Criteria:

* Ages18 to 34
* Smoke little cigars/cigarillos (LCCs) "some days" or "everyday"
* Ability to read English at an 8th grade level or higher
* No immediate plans to quit using tobacco

Exclusion Criteria:

* Current use of nicotine replacement therapy (NRT)
* Pregnant, planning to become pregnant, or currently breastfeeding
* Past or current self-reported clinically significant heart disease or hypertension, or other smoking-related disease (by history) that preclude successful study completion Inability to abstain from nicotine/tobacco products for at least 12 hours prior to each of two study sessions
* Report using the study cigarillo brand as their preferred brand (as this will likely unduly influence their perceptions)
* Unwillingness to use "untipped" (e.g., plastic or wood tip) little cigars/cigarillos.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Subjective response to smoking | Laboratory visits, up to 3 weeks after the baseline
  average ratings of psychological reward following smoking from Modified Cigarette Evaluation Scale. Higher scores indicate higher reward. Score responses range from 1 to 7
Number of cigarillos smoked | Daily smartphone surveys, up to 3 weeks after the baseline
  The number of cigarillos smoked during each 7-day take-home period

CONTACTS AND LOCATIONS:
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Sharing may be available at the discretion and with the permission of the university and an approved data use agreement.